CLINICAL TRIAL: NCT04397913
Title: Population Pharmacokinetics and Dosage Individualization of Paracetamol and Ibuprofen in Preterm Neonates and Infants With Patent Ductus Arteriosus
Brief Title: Population Pharmacokinetics and Dosage Individualization of Paracetamol and Ibuprofen in Children With PDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhao, Professor; Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: 2020paracetamol-ibuprofen001
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment(paracetamol or ibuprofen): Paracetamol and ibuprofen are administered at standard dose for children with PDA.
  Interventions: Drug: Paracetamol; Drug: Ibuprofen

INTERVENTIONS:
Drug: Paracetamol — 15 mg/kg, q6h
  Other Names: Acetaminophen
Drug: Ibuprofen — 10 mg/kg qd for the 1st day, 5 mg/kg qd for the 2nd and 3rd day

SUMMARY:
The investigator's purpose is to study the population pharmacokinetics of paracatamol and ibuprofen in neonates with patent ductus arteriosus (PDA) and assess the feasibility of dosage individualization.

DETAILED DESCRIPTION:
The investigator's purpose is to study the population pharmacokinetics of paracatamol and ibuprofen in neonates with patent ductus arteriosus (PDA) and assess the feasibility of dosage individualization. In this study, the investigator will detect drug concentration in plasma and other clinical test to construct population pharmacokinetic models.

ELIGIBILITY:
Inclusion Criteria:

* Patients have been diagnosed with PDA;
* Age: postnatal age ≤ 28 days;
* Paracetamol or ibuprofen used as part of regular treatment;
* Paracetamol or ibuprofen was administered orally.

Exclusion Criteria:

* Patients who die within the treatment cycle;
* Patients with other heart diseases;
* Other factors that the researcher considers unsuitable for inclusion.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with patent ductus arteriosus
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-25 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-05-06 (Estimated)

PRIMARY OUTCOMES:
Plasma drug concentration of paracetamol | at (0-1) hour, (1-3) hours, (3-5) hours, (5-6) hours after oral administration
  To detect the plasma concentration of paracetamol after administration
Plasma drug concentration of ibuprofen | at (0-1.5) hours, (1-4) hours, (4-12) hours,(12-24) hours after oral administration
  To detect the plasma concentration of ibuprofen after administration
Echocardiography | Through study completion, an average of 3 days
  To measure arterial duct diameter, shunt speed and direction of shunt
Cardiac function | Through study completion, an average of 3 days
  To detect brain natriuretic peptide(BNP) and troponin T(cTnT)

SECONDARY OUTCOMES:
Adverse events | Through study completion, an average of 3 days
  Drug-related adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Chengdu, Sichuan, China